CLINICAL TRIAL: NCT05775939
Title: PET Functional Imaging to Evaluate Cardiac Radiation Damage (EUCLID)
Brief Title: PET/CT Imaging to Evaluate Cardiac Radiation Damage in Patients With Lung or Esophageal Cancer, EUCLID Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22D.705; JT 20888 (Other: JeffTrial Number)
Record Dates: First submitted 2023-02-07; First posted 2023-03-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Carcinoma; Esophageal Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (sarcoidosis FDG PET-CT) (Experimental): Patients undergo sarcoidosis FDG PET-CT of the heart before, during and, after radiotherapy.
  Interventions: Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Other: Fludeoxyglucose F-18 — Given FDG
  Other Names: 105851-17-0; 18FDG; 2-Deoxy-2-(18F)Fluoro-D-Glucose; 2-F18-Fluoro-2-deoxy-D-glucose; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging; PET; PET SCAN; Positron Emission Tomography Scan; proton magnetic resonance spectroscopic imaging; Positron-Emission Tomography; PT
Procedure: Computed Tomography — Undergo PET-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial examines positron emission tomography (PET)/computed tomography (CT) in evaluating cardiac radiation damage in patients with lung or esophageal cancer. As part of the treatment for lung or esophageal cancer, patients will undergo radiation therapy. Sometimes, during this treatment, the heart is also subjected to some radiation which could affect its function, either increasing or decreasing the function. It is not known the consequences of this change nor is it known if doctors can detect the changes associated with the radiation. Sarcoidosis FDG positron emission tomography (PET)-computed tomography (CT) scans are a common way to image cardiac inflammation and myocardial viability. This study may help doctors image the heart before, during and after radiotherapy to monitor any changes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize radiation-related functional imaging changes in the heart using sarcoidosis fludeoxyglucose F-18 (FDG) PET-CT imaging.

SECONDARY OBJECTIVES:

I. 1. To evaluate the ability of imaging changes in the heart to predict for overall survival (OS).

II. To evaluate the ability of imaging changes in the heart to predict for cardiac toxicity.

III. To evaluate the ability of imaging changes in the heart to predict for cardiac related death.

EXPLORATORY OBJECTIVES:

I. To evaluate radiation treatment planning strategies to reduce risk of cardiotoxicity.

II. To determine the correlation between sarcoidosis FDG PET-CT scans and oncologic FDG PET-CT scans.

OUTLINE:

Patients undergo sarcoidosis FDG PET-CT of the heart before, during and, after radiotherapy.

After completion of study treatment, patients are followed up at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged >= 18
* Life expectancy >= 3 months as assessed by Radiation Oncologist
* Mean heart dose estimated by Radiation Oncologist to be >= 5 Gy (physics dose or biologically equivalent dose)
* Pathologically proven (either histologic or cytologic) proven lung cancer or esophageal cancer
* Planned radiation treatment course for management of lung or esophageal cancer * Both standard and hypofractionation schedules are permitted

Exclusion Criteria:

* Contraindication for FDG PET-CT scans as assessed by the radiation oncologist or nuclear medicine radiologist
* Palliative radiation doses defined as 20 Gy in 5 fractions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean standardized uptake value (SUV) changes in the heart | Up to 30 months after radiotherapy
  Measured by sarcoidosis fludeoxyglucose F-18 (FDG) positron emission tomography (PET)-computed tomography (CT) scans.

SECONDARY OUTCOMES:
Ability of pre- to post-radiotherapy SUV changes in the heart | Up to 30 months after radiotherapy
  Measured by sarcoidosis FDG PET-CT scans.
Overall survival | Up to 30 months after radiotherapy
  Survival
Cardiac toxicity | Up to 30 months after radiotherapy
  Assessed using >= grade 2 and >= grade cardiac events using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Cardiac toxicity judged to be secondary to radiotherapy by cardiologist and radiation oncologist | Up to 30 months after radiotherapy
  Judged to be secondary to radiotherapy by cardiologist and radiation oncologist
Cardiac related death | Up to 30 months after radiotherapy
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Yevgeniy Vinogradskiy, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States